CLINICAL TRIAL: NCT06265584
Title: Phase II Clinical Trial of 2 Step ATG Combined With Tacrolimus and Mini Methotrexate for Prevention of Acute GVHD Post Reduced Intensity Allogeneic Stem Cell Transplant
Brief Title: Trial of 2 Step ATG for Prevention of Acute GVHD Post Allogeneic Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300011730 (UAB2370); Robert Award (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Acute Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorders
Keywords: Leukemia; Myelodysplastic Syndrome; Myeloproliferative
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- phase II single arm study of 2 step ATG dosing in prevention of aGVHD (Experimental): The primary outcome for the study is GRFS rate at one-year post transplant. GRFS will be estimated using Kaplan Meier method The reported GRFS with recent phase III trial of PTCY/tac/MMF in transplant from matched related and unrelated donors at 1 year follow up was 52%. We hypothesize that with 2 step ATG/Tac/Mini MTX regimen, we can achieve a one year GRFS of 69%.
  Interventions: Drug: ATG dosing platform when combined with standard tacrolimus and mini methotrexate

INTERVENTIONS:
Drug: ATG dosing platform when combined with standard tacrolimus and mini methotrexate — On Day -8, you will be admitted to the hospital and receive a dose of prednisone at 1 mg/kg (ATG premedication). You will receive a steroids 3 hours before every ATG infusion. On day -7, you will receive a small dose of ATG as an intravenous (IV) infusion. ATG will be repeated on days -6, -5 and -1. Routine transplant chemotherapy agent fludarabine will be given on days -7 to -3 as daily IV infusions. Melphalan, another routine transplant chemotherapy will be given on day -4 as IV infusion. Tacrolimus (standard immune suppression agent) will start on day -3 as continuous IV infusion and switched to oral after engraftment. Methotrexate is another standard immune suppression medication which is given IV on day +1, +3, +6, and +11 post-transplant. We plan to draw blood on days -4,, -1, +3, +7, and +14 to measure ATG levels.

SUMMARY:
In an effort to reduce graft versus host disease (GVHD) and enhance graft versus leukemia (GVL) effect post allogenic hematopoietic stem cell transplantation (AHSCT), recent research has focused on host immune cell depletion. Frame shifting anti-thymocyte globulin (ATG) backwards to earlier days before days 0 can result in deeper host and less graft T-cell depletion, leading to better immune reconstitution. Preliminary data where 80% of the ATG dose is given on days -6,-5,-4 and 20% given on day -1, showed effective prevention of severe acute GVHD, chronic GVHD and favorable early immune reconstitution. We hypothesize that our 2 step ATG dosing platform when combined with standard tacrolimus and mini methotrexate can prevent grade III-IV acute GVHD and chronic GVHD, resulting in improvement of GVHD/relapse free survival at one year post transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, age 18-75 years
2. Patients must have a related or unrelated peripheral blood stem cell donor. Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation. Unrelated donor must be 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be willing to donate peripheral blood stem cells and be medically eligible to donate stem cells according to NMDP criteria.
3. A candidate for reduced intensity preparative regimen, based on age≥60, or HCT-CI of ≥4, or considered by the treating physician to have high risk for toxicity with myeloablative preparative regimen.
4. Cardiac function: Ejection fraction >40%
5. Measured creatinine clearance greater than 50 mL/minute (using the Cockcroft-Gault formula and actual body weight)
6. Pulmonary function: DLCO ≥50% (adjusted for hemoglobin) and FEV1≥50%
7. Liver function: total bilirubin < 1.5x the upper limit of normal and ALT/AST < 2.5x the upper normal limit. Patients who have been diagnosed with Gilbert's Disease are allowed to exceed the defined bilirubin value of up to <3mg/dl.
8. Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two effective methods of contraception or agree to complete abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
9. Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
10. Karnofsky performance status KPS ≥ 70
11. Patients must have a diagnosis of one of the following:

    A-AML with either detectable AML on pre AHSCT bone marrow (microscopic ≤5, flow or cytogenetic), or adverse cytogenetic, or molecular features (≥ 4 clonal abnormalities, or monosomal karyotype, inv(3)/t(3;3) or, EV11+, FLT3-ITD (+) without MPN1, P53 mutation positive, ASXL1+, mutant RUNX1.

    B- MDS with the following features: Residual blasts > 5% blasts in the bone marrow after hypomethylating agents +/- venetoclax, MDS with high IPSS-R and monosomal karyotype, MDS with P-53 or JAK2 mutation.

    C-Myelofibrosis with blasts in the peripheral blood.
12. The subject is willing and able to signed informed consent and abide by the protocol requirements.

Exclusion Criteria:

1. Autologous hematopoietic stem cell transplant < 3 months prior to enrollment.
2. Patients with florid residual AML with > 5% blast in the marrow or circulating blast in the peripheral blood are not eligible for this study.
3. Previous allogeneic stem cell transplant.
4. Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
5. Known hypersensitivity to one or more of the study agents
6. Received any investigational drugs within the 14 days prior to the first day of transplant conditioning
7. Pregnant and/or breastfeeding
8. Evidence of HIV infection or known HIV positive serology.
9. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
10. Patient with documented cirrhosis
11. Non-hematologic malignancy within prior three (3) years, with the exception of squamous cell or basal cell skin carcinoma. Patients with prior malignancies except resected localized non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the PI
12. Participation in another clinical study with an investigational product during the last 28 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Rate of GRFS (graft versus host disease GVHD, relapse free survival) at one year post transplant. | 1 year post transplant
  Rate of GRFS is defined as the time from date of first dose of fludarabine until occurrence of grade III-IV aGVHD, and or cGVHD requiring systemic immune suppression, and or disease progression or death whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al Kadhimi, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States